CLINICAL TRIAL: NCT05920083
Title: Noctural Pulse Waves Variations in OSA as a Predictor of Autonomic and Vascular Response to CPAP Therapy
Brief Title: Obstructive Sleep Apnea - Autonomic and Vascular Exploration
Acronym: OSAVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting desired number of participant.
Sponsor: Raphael Heinzer (Other)
Responsible Party: Sponsor-Investigator, Raphael Heinzer, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01012023
Record Dates: First submitted 2023-06-06; First posted 2023-06-27 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: one group, before-after design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPAP withdrawal (Experimental): CPAP withdrawal for 2 weeks
  Interventions: Other: CPAP withdrawal

INTERVENTIONS:
Other: CPAP withdrawal — 2 weeks of CPAP withdrawal

SUMMARY:
The goal of this clinical trial is to assess the effect of CPAP withdrawal on vascular and autonomic function in patients with obstructive sleep apnea. The main question it aims to answer is:

• Is the pulse wave amplitude index able to predict the impact of sleep apnea treatment withdrawal (continuous positive airway pressure, CPAP) on endothelial function and baroreflex sensitivity?

Participants will stop using their CPAP for 2 weeks and the investigators will assess vascular and autonomic function before and after the withdrawal. Researchers will compare endothelial and autonomic function at baseline and after 2 weeks of withdrawal to see if there are differences. Moreover, they will assess the association between pulse wave amplitude drop profile and effect of CPAP withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Diagnosed with OSA (AHI ≥15 events/h), confirmed during screening period
* Adequately treated with CPAP therapy for ≥6 months
* Able to give informed consent as documented by signature

Exclusion Criteria:

* Professional drivers will be excluded from the study because temporary withdrawal of CPAP may induce drowsiness.
* We will also exclude patients with conditions that may affect endothelial and autonomic function:

  * Known Diabetes
  * Known heart failure
  * Known chronic kidney disease
  * Pregnant or lactating women
  * Morbid obesity (≥40 kg/m2)
  * Known Excessive alcohol consumption
  * Known Dementia (especially dementia with Lewy bodies). (61)
  * Patients using alpha and beta blockers
  * Known atrial fibrillation
  * Inability to follow the procedures of the study due to language problems or psychological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Change in flow-mediated dilation | Between FMD measured after 2 weeks of CPAP withdrawal and FMD measured after 2 weeks on CPAP
  Endothelial function as measured with flow-mediated dilation
Change in the slope of baroreflex sensitivity | Between BRS measured after 2 weeks of CPAP withdrawal and BRS measured after 2 weeks on CPAP
  Autonomic function as measure with the slope of BRS

SECONDARY OUTCOMES:
Arterial stiffness assessed by the pulse transit time | Baseline, after 2 weeks of withdrawal, after 2 weeks on CPAP
  arterial stiffness measured by the pulse transit time
Nocturnal heart rate variability indices (linear and non linear) | baseline, after 2 weeks of withdrawal, after 2 weeks on CPAP
  HRV measured on the ECG of polygraphy
Change in heart rate response to the cold pressure test | baseline, after 2 weeks of withdrawal, after 2 weeks on CPAP
  delta heart rate before and after cold pressure test
Hypoxic burden | baseline, after 2 weeks of withdrawal, after 2 weeks on CPAP
  hypoxic burden of sleep apnea based on polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Heinzer, Pr., Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV)
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No